CLINICAL TRIAL: NCT00703014
Title: Pregnancy and Neonatal Follow-up of Ongoing Pregnancies Established After Controlled Ovarian Stimulation in Clinical Trial 38819 for Org 36286 (Corifollitropin Alfa)
Brief Title: Pregnancy and Neonatal Follow-up of Ongoing Pregnancies Established in Clinical Trial P05787 (P05712)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: P05712; 2004-004772-36 (EudraCT Number); 38821 (Other: Organon); MK-8962-005 (Other: Merck)
Record Dates: First submitted 2008-06-18; First posted 2008-06-20 (Estimated); Results first posted 2014-11-24 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2022-02

CONDITIONS: Pregnancy; Neonates
Keywords: Neonatal outcome; Congenital malformations; In-Vitro fertilization; Controlled ovarian stimulation; Follow-up
MeSH Terms: conditions — Congenital Abnormalities | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide; follitropin beta; ganirelix; Progesterone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Mothers Corifollitropin Alfa 150 µg: Participants from the Base Trial P05787 who received a single subcutaneous (SC) injection of 150 µg Corifollitropin Alfa on day 2 or 3 of the menstrual cycle (Stimulation Day 1); 7 daily SC injections from Stimulation Days 1 to 7 with placebo-recombinant Follicle Stimulating Hormone (recFSH); followed by daily SC injections with 200 IU recFSH up to the day of human chorionogonadotropin (hCG); multiple daily SC injections of Ganirelix from Stimulation Day 5 to the day of hCG; a single dose of hCG (5000 or 10,000 IU/USP) was administered when 3 follicles >= 17 mm were observed; and on the day of oocyte pick up (OPU) daily doses of progesterone were started and continued for up to 6 weeks or menses. Eligible participants from the Base Trial were enrolled in Follow Up Trial P05712, where no study treatments were given, and pregnancy, delivery and neonatal outcome were monitored.
  Interventions: Drug: Corifollitropin Alfa 150 μg; Drug: Placebo for RecFSH/Follitropin beta; Biological: 200 IU RecFSH/Follitropin beta (Days 8 to hCG); Drug: Ganirelix; Biological: hCG; Biological: Progesterone
- Mothers recFSH 200 IU: Participants from the Base Trial P05787 who received a single SC injection of placebo Corifollitropin Alfa on day 2 or 3 of the menstrual cycle (Stimulation Day 1); 7 daily SC injections with 200 IU recFSH from Stimulation Days 1 to 7; followed by daily SC injections with 200 IU recFSH up to the day of hCG; multiple daily SC injections of Ganirelix from Stimulation Day 5 to the day of hCG; a single dose of hCG (5000 or 10,000 IU/USP) was administered when 3 follicles >= 17 mm were observed; and on the day of OPU daily doses of progesterone were started and continued for up to 6 weeks or menses. Eligible participants from the Base Trial were enrolled in Follow Up Trial P05712, where no study treatments were given, and pregnancy, delivery and neonatal outcome were monitored.
  Interventions: Biological: 200 IU RecFSH/Follitropin beta (Days 1 to 7); Drug: Placebo for Corifollitropin Alfa; Biological: 200 IU RecFSH/Follitropin beta (Days 8 to hCG); Drug: Ganirelix; Biological: hCG; Biological: Progesterone

INTERVENTIONS:
Drug: Corifollitropin Alfa 150 μg — In the Base Trial P05787, on the morning of day 2 or 3 of the menstrual cycle (Stimulation Day 1), a single SC injection of 150 μg (0.5 mL) Corifollitropin Alfa was administered in the abdominal wall.
  Groups: Mothers Corifollitropin Alfa 150 µg
Biological: 200 IU RecFSH/Follitropin beta (Days 1 to 7) — In the Base Trial P05787, daily SC injections with 200 IU fixed dose recFSH were started on Stimulation Day 1 and continued up to and including Stimulation Day 7.
  Other Names: follitropin beta; Puregon®; Follistim®
  Groups: Mothers recFSH 200 IU
Drug: Placebo for Corifollitropin Alfa — In the Base Trial P05787, on the morning of day 2 or 3 of the menstrual cycle (Stimulation Day 1), a single SC injection from a pre-filled syringe containing an identical solution when compared to Corifollitropin Alfa was administered in the abdominal wall.
  Groups: Mothers recFSH 200 IU
Drug: Placebo for RecFSH/Follitropin beta — In the Base Trial P05787, daily SC injections of an identical ready-for-use solution, but without the active ingredient, supplied in cartridges for SC injection with the Follistim Pen, were started on Stimulation Day 1 and continued up to and including Stimulation Day 7.
  Groups: Mothers Corifollitropin Alfa 150 µg
Biological: 200 IU RecFSH/Follitropin beta (Days 8 to hCG) — In the Base Trial P05787, from Stimulation Day 8 onwards a daily SC dose of 200 IU recFSH was administered up to and including the Day of hCG.
Drug: Ganirelix — In the Base Trial P05787, on Stimulation Day 5 a daily SC injection of 0.25 mg was started, which continued up to and including the day of hCG.
Biological: hCG — In the Base Trial P05787, when 3 follicles >= 17 mm were observed by USS, a single dose of 10,000 IU/USP hCG was administered; or, for those at risk for Ovarian Hyperstimulation Syndrome (OHSS), a lower dose of 5,000 IU/USP
Biological: Progesterone — In the Base Trial P05787, on the day of OPU, luteal phase support was started by administering micronized progesterone of at least 600 mg/day vaginally, or at least 50 mg/day intramuscular (IM), which continued for at least 6 weeks, or up to menses.

SUMMARY:
The objective of this trial was to evaluate whether Corifollitropin Alfa treatment for the induction of multifollicular growth in women undergoing controlled ovarian stimulation (COS) prior to in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI) was safe for pregnant participants and their offspring. The primary endpoint was the take-home baby rate calculated as the number of participants with an ongoing pregnancy in Base Trial P05787 (NCT00696800) with at least one live born infant relative to the number of participants in the Base Trial, and to the number of participants in the Base Trial with Embryo Transfer (ET).

DETAILED DESCRIPTION:
This is a follow-up protocol to prospectively monitor pregnancy, delivery, and neonatal outcome of all women who were treated with Corifollitropin Alfa or recFSH and became pregnant during Base Trial P05787 (NCT00696800). For this trial, no study specific assessments are required, but information as obtained in standard practice will be used.

ELIGIBILITY:
Inclusion Criteria:

* Participants who received at least one dose of either Corifollitropin Alfa or

Puregon®/Follistim® AQ Cartridge in Base Trial P05787 (NCT00696800);

* Ongoing pregnancy confirmed by ultrasound at least 10 weeks after embryo transfer in Base Trial P05787 (NCT00696800);
* Able and willing to give written informed consent.

Exclusion Criteria:

* None

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with an ongoing pregnancy at least 10 weeks after ET in Base Trial P05787 (NCT00696800) were enrolled in this trial.
Sampling Method: Non-Probability Sample
Enrollment: 541 (Actual)
Dates: Start 2006-07-13 (Actual); Primary Completion 2008-04-18 (Actual); Study Completion 2009-03-15 (Actual)

REFERENCES:
- [Derived] Bonduelle M, Mannaerts B, Leader A, Bergh C, Passier D, Devroey P. Prospective follow-up of 838 fetuses conceived after ovarian stimulation with corifollitropin alfa: comparative and overall neonatal outcome. Hum Reprod. 2012 Jul;27(7):2177-85. doi: 10.1093/humrep/des156. Epub 2012 May 15. PMID 22587997
- [Derived] Boostanfar R, Mannaerts B, Pang S, Fernandez-Sanchez M, Witjes H, Devroey P; Engage Investigators. A comparison of live birth rates and cumulative ongoing pregnancy rates between Europe and North America after ovarian stimulation with corifollitropin alfa or recombinant follicle-stimulating hormone. Fertil Steril. 2012 Jun;97(6):1351-8. doi: 10.1016/j.fertnstert.2012.02.038. Epub 2012 Mar 28. PMID 22459628

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Period one consists of mothers from the Base Trial P05787 (NCT00696800), randomized to treatment groups Corifollitropin Alfa (Org 36286) or recombinant Follicle Stimulating Hormone (recFSH). Period two consists of mothers (N = 541) who enrolled in trial P05712. Period three consists of miscarried/stillborn fetuses and infants born in trial P05712.
Groups:
- Mothers Corifollitropin Alfa 150 µg: Participants from the Base Trial P05787 (NCT00696800) who received a subcutaneous (SC) injection of 150 µg Corifollitropin Alfa on day 2 or 3 of the menstrual cycle (Stimulation Day 1); 7 daily SC injections from Stimulation Days 1 to 7 with placebo-recFSH; followed by daily SC injections with 200 IU recFSH up to the day of human Chorion Gonadotropin (hCG); multiple daily SC injections of Ganirelix from Stimulation Day 5 to the day of hCG; a single dose of hCG (10,000 or 5,000 IU/USP) was administered when 3 follicles >= 17 mm were observed; and on the day of oocyte pick-up (OPU) daily doses of progesterone were started and continued for up to 6 weeks or menses. Eligible participants from the Base Trial were enrolled in Follow Up Trial P05712, where no study treatments were given, and pregnancy, delivery and neonatal outcome were monitored.
- Mothers recFSH 200 IU: Participants from the Base Trial P05787 (NCT00696800) who received a single SC injection of placebo Corifollitropin Alfa on day 2 or 3 of the menstrual cycle (Stimulation Day 1); 7 daily SC injections with 200 IU recFSH from Stimulation Days 1 to 7; followed by daily SC injections with 200 IU recFSH up to the day of hCG; multiple daily SC injections of Ganirelix from Stimulation Day 5 to the day of hCG; single dose of hCG (10,000 or 5,000 IU/USP) was administered when 3 follicles >= 17 mm were observed; and on the day of OPU daily doses of progesterone were started and continued for up to 6 weeks or menses. Eligible participants from the Base Trial were enrolled in Follow Up Trial P05712, where no study treatments were given, and pregnancy, delivery and neonatal outcome were monitored.
- Fetuses/Infants Corifollitropin Alfa 150 µg: Fetuses and infants born in Follow Up Trial P05712 to mothers treated with Corifollitropin Alfa 150 µg in Base Trial P05787 (NCT00696800)
- Fetuses/Infants recFSH 200 IU: Fetuses and infants born in Follow Up Trial P05712 to mothers treated with recFSH 200 IU in Base Trial P05787 (NCT00696800)
Period: Mothers Base Trial P05787 (NCT00696800)
Arm/Group | Mothers Corifollitropin Alfa 150 µg | Mothers recFSH 200 IU | Fetuses/Infants Corifollitropin Alfa 150 µg | Fetuses/Infants recFSH 200 IU
Started | 757 (Randomized in Base Trial P05787 (NCT00696800)) | 752 (Randomized in Base Trial P05787 (NCT00696800)) | 0 | 0
Treated | 756 (Intent-To-Treat (ITT) group in Base Trial P05787 (NCT00696800)) | 750 (ITT group in Base Trial P05787 (NCT006968000)) | 0 | 0
Embryo Transfer | 672 (Embryo transfer (ET) in Base Trial P05787 (NCT006968000)) | 704 (Embryo transfer (ET) in Base Trial P05787 (NCT006968000)) | 0 | 0
Completed | 295 (ITT group in P05712, ongoing pregnancy at 10 weeks after ET in Base Trial P05787 (NCT006968000)) | 286 (ITT group in P05712, ongoing pregnancy at 10 weeks after ET in Base Trial P05787 (NCT006968000)) | 0 | 0
Not Completed | 462 | 466 | 0 | 0
Period: Mothers Follow Up Trial P05712
Arm/Group | Mothers Corifollitropin Alfa 150 µg | Mothers recFSH 200 IU | Fetuses/Infants Corifollitropin Alfa 150 µg | Fetuses/Infants recFSH 200 IU
Started | 274 (Eligible participants who completed Base Trial P05787 and then enrolled in Follow Up Trial P05712) | 267 (Eligible participants who completed Base Trial P05787 and then enrolled in Follow Up Trial P05712) | 0 | 0
Completed | 241 (Completed Follow Up in Trial P05712) | 235 (Completed Follow Up in Trial P05712) | 0 | 0
Not Completed | 33 | 32 | 0 | 0
Not completed — Did not complete follow up in P05712 | 33 | 32 | 0 | 0
Period: Fetuses/Infants Follow Up Trial P05712
Arm/Group | Mothers Corifollitropin Alfa 150 µg | Mothers recFSH 200 IU | Fetuses/Infants Corifollitropin Alfa 150 µg | Fetuses/Infants recFSH 200 IU
Started | 0 | 0 | 352 (Fetuses in Follow Up Trial P05712) | 326 (Fetuses in Follow Up Trial P05712)
Live Born Infants | 0 | 0 | 344 (Live born infants in Follow Up Trail P05712) | 315 (Live born infants in Follow Up Trail P05712)
Completed | 0 | 0 | 305 (Infants in P05712 with Follow Up Completed) | 284 (Infants in P05712 with Follow Up Completed)
Not Completed | 0 | 0 | 47 | 42
Not completed — Did not complete follow up in P05712 | 0 | 0 | 47 | 42

BASELINE CHARACTERISTICS:
Population: Eligible mothers from the Base Trial P05787 (NCT00696800) who enrolled in Follow Up Trial P05712
Groups:
- Mothers Corifollitropin Alfa 150 µg: Participants from the Base Trial P05787 (NCT00696800) who received a SC injection of 150 µg Corifollitropin Alfa on day 2 or 3 of the menstrual cycle (Stimulation Day 1); 7 daily SC injections from Stimulation Days 1 to 7 with placebo-recFSH; followed by daily SC injections with 200 IU recFSH up to the day of hCG; multiple daily SC injections of Ganirelix from Stimulation Day 5 to the day of hCG; a single dose of hCG (10,000 or 5,000 IU/USP) was administered when 3 follicles >= 17 mm were observed; and on the day of OPU daily doses of progesterone were started and continued for up to 6 weeks or menses. Eligible participants from the Base Trial were enrolled in Follow Up Trial P05712, where no study treatments were given, and pregnancy, delivery and neonatal outcome were monitored.
- Total: Total of all reporting groups
Arm/Group | Mothers Corifollitropin Alfa 150 µg | Mothers recFSH 200 IU | Total
Number analyzed (Participants) | 274 | 267 | 541
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.4 (3.2) | 31.3 (3.5) | 31.3 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 274 | 267 | 541
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Mothers in Current Follow Up Trial Experiencing Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a trial participant administered a pharmaceutical product, and which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including laboratory finding), symptom, or disease temporally associated with the use of investigational medicinal product.
Time Frame: Up to one day following delivery (up to 1 year)
Population: Eligible Mothers from the Base Trial P05787 (NCT00696800) who enrolled in the Follow Up Trial P05712. Infants from Follow Up Trial P05712 were not analyzed in this outcome measure.
Measure: Number; unit: Participants
Arm/Group | Mothers Corifollitropin Alfa 150 µg | Mothers recFSH 200 IU
Number analyzed (Participants) | 274 | 267
Participants | 222 | 214

2. Primary Outcome: Number of Mothers in Current Follow Up Trial Experiencing Serious AEs (SAEs)
Description: A SAE is any untoward medical occurrence that at any dose resulted in the following: death, was life threatening, required in-patient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, or was a congenital anomaly/birth defect.
Time Frame: Up to one day following delivery (up to 1 year)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Mothers Corifollitropin Alfa 150 µg | Mothers recFSH 200 IU
Number analyzed (Participants) | 274 | 267
Participants | 129 | 117

3. Primary Outcome: Number of Infants Born in Current Follow Up Trial Experiencing AEs
Description: as for outcome 1
Time Frame: Up to 12 weeks following delivery (up to 1 year)
Population: Infants born in Follow Up Trial P05712. Mothers were not analyzed in this outcome measure.
Measure: Number; unit: Participants
Groups:
- Infants Corifollitropin Alfa 150 µg: Infants born in Follow Up Trial P05712 to mothers treated with Corifollitropin Alfa 150 µg in Base Trial P05787 (NCT00696800)
- Infants recFSH 200 IU: Infants born in Follow Up Trial P05712 to mothers treated with recFSH 200 IU in Base Trial P05787 (NCT00696800)
Arm/Group | Infants Corifollitropin Alfa 150 µg | Infants recFSH 200 IU
Number analyzed (Participants) | 344 | 315
Participants | 164 | 161

4. Primary Outcome: Number of Infants in Current Follow Up Trial Experiencing SAEs
Description: as for outcome 2
Time Frame: Up to 12 weeks following delivery (up to 1 year)
Population: Infants born in Follow Up Trial P05712. Mothers were not analyzed in this outcome measure.
Measure: Number; unit: Participants
Arm/Group | Infants Corifollitropin Alfa 150 µg | Infants recFSH 200 IU
Number analyzed (Participants) | 344 | 315
Participants | 106 | 94

5. Primary Outcome: Percentage of Mothers From the Base Trial P05787 With at Least One Live Born Infant (Take-home Baby Rate) Relative to the Number of Participants in the Base Trial.
Description: The take-home baby rate is 100 X the number of participants with an ongoing pregnancy in Base Trial P05787 (NCT00696800), from the Intent-to-Treat (ITT) group, with at least one live born infant relative to the number of participants in the Base Trial.
Time Frame: At least 10 weeks after embryo transfer in Base Trial P05787 up to birth in current follow up Trial (up to 1 year)
Population: Mothers from the ITT group of the Base Trial P05787 (NCT00696800). Infants from Follow Up Trial P05712 were not analyzed in this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Mothers Corifollitropin Alfa 150 µg | Mothers recFSH 200 IU
Number analyzed (Participants) | 756 | 750
Percentage of Participants | 35.6 | 34.4

6. Primary Outcome: Percentage of Mothers From the Base Trial P05787 With at Least One Live Born Infant (Take-home Baby Rate) Relative to the Number of Participants From the Base Trial With Embryo Transfer.
Description: The take-home baby rate is 100 X the number of participants with an ongoing pregnancy in Base Trial P05787 (NCT00696800), from the ITT group, with at least one live born infant relative to the number of participants from the Base Trial with embryo transfer.
Time Frame: At least 10 weeks after embryo transfer in Base Trial P05787 up to birth in current Follow Up Trial (up to 1 year)
Population: Mothers from the ITT group of the Base Trial P05787 (NCT00696800) who had ET. Infants from Follow Up Trial P05712 were not analyzed in this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Mothers Corifollitropin Alfa 150 µg | Mothers recFSH 200 IU
Number analyzed (Participants) | 672 | 704
Percentage of Participants | 40.0 | 36.6

ADVERSE EVENTS:
Time Frame: Mothers: up to one day after delivery; Fetuses and Infants: up to 12 weeks after birth
Description: All study treatments were considered to be administered to the mother.
Arm/Group | Mothers Corifollitropin Alfa 150 µg | Mothers recFSH 200 IU | Fetuses/Infants Corifollitropin Alfa 150 µg | Fetuses/Infants recFSH 200 IU
Serious Adverse Events (participants affected / at risk) | 129/274 | 117/267 | 106/352 | 94/326
Other Adverse Events (participants affected / at risk) | 112/274 | 118/267 | 37/352 | 41/326
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mothers Corifollitropin Alfa 150 µg (N=274) | Mothers recFSH 200 IU (N=267) | Fetuses/Infants Corifollitropin Alfa 150 µg (N=352) | Fetuses/Infants recFSH 200 IU (N=326)
Anaemia neonatal (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 6 (6) | 3 (3)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Placental transfusion syndrome (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia neonatal (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bradycardia foetal (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bradycardia neonatal (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest neonatal (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nodal rhythm (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia foetal (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Abnormal palmar/planta creases (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Accessory auricle (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 5 (5) | 11 (11)
Atrioventricular septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bat ear (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cervical rib (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chondrodystrophy (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cleft lip (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cleft palate (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Cleft uvula (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clinodactyly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital anaemia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital aortic anomaly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital aortic stenosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital aortic valve stenosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital central nervous system anomaly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Congenital cerebral cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital choroid plexus cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Congenital coronary artery malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congenital cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congenital eyelid malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Congenital foot malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congenital hand malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congenital hearing disorder (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital hip deformity (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Congenital hydrocephalus (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Congenital inguinal hernia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital labia pudendi adhesions (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congenital mitral valve stenosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital naevus (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Congenital nose malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congenital optic nerve anomaly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital ovarian anomaly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congenital pyelocaliectasis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Congenital spinal cord anomaly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital torticollis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congenital tracheomalacia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Craniotabes (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cryptorchism (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
Duodenal atresia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Exomphalos (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 7 (7) | 3 (3)
Eyelid ptosis congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fallot's tetralogy (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemangioma congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
Heart disease congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip dysplasia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Hypertelorism of orbit (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypospadias (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Immunodeficiency congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 5 (5) | 6 (6)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pilonidal cyst congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Plagiocephaly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pulmonary artery stenosis congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pulmonary valve stenosis congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Rhesus haemolytic disease of newborn (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Single umbilical artery (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skull malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Strabismus congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supernumerary nipple (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syndactyly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Talipes (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Trisomy 21 (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Secondary hypogonadism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Eye disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacrimal cyst (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinopathy of prematurity (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Anal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Necrotising enterocolitis neonatal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Short-bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug withdrawal syndrome neonatal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever neonatal (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal multi-organ faillure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sudden infant death syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 9 (9) | 8 (8)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neonatal cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Genital herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incision site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neonatal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neonatal pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis neonatal (Infections and infestations) | 0 (0) | 0 (0) | 7 (7) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acoustic stimulation tests abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Amniotic fluid volume decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose fluctuation (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood sodium increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Body temperature decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 6 (6) | 3 (3)
Cytomegalovirus antibody positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foetal heart rate abnormal (Investigations) | 3 (3) | 2 (2) | 2 (2) | 0 (0)
Foetal heart rate decreased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Haemoglobin Barts present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heart rate decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cow's milk intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatty acid deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gestational diabetes (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia neonatal (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Loctose intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotonia neonatal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Positional plagiocephaly (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Posture abnormal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage neonatal (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral ventricle dilatation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Convulsion neonatal (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy neonatal (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intraventricular haemorrhage neonatal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neurological symptom (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Superior sagittal sinus thrombosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Antepartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arrested labour (Pregnancy, puerperium and perinatal conditions) | 12 (12) | 15 (15) | 0 (0) | 0 (0)
Breech presentation (Pregnancy, puerperium and perinatal conditions) | 26 (26) | 23 (23) | 0 (0) | 0 (0)
Caput succedaneum (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 3 (3) | 0 (0) | 0 (0)
Cervical incompetence (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Chorioamnionitis (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Discordant twin (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Face presentation (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Failed induction of labour (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 6 (6) | 13 (13) | 1 (1) | 2 (2)
Foetal growth retardation (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Foetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foetal macrosomia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foetal malposition (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foetal malpresentation (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 4 (4) | 0 (0) | 0 (0)
HELLP syndrome (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hydrops foetalis (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Imminent abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intrapartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 8 (8) | 8 (8)
Meconium in amniotic fluid (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Meconium stain (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Multiple pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Placenta accreta (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Placenta praevia (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 12 (12) | 10 (10) | 0 (0) | 0 (0)
Pregnancy induced hypertension (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 56 (56) | 48 (48)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 37 (37) | 33 (33) | 0 (0) | 0 (0)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 8 (8) | 6 (6) | 0 (0) | 0 (0)
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 6 (6) | 1 (1) | 0 (0) | 0 (0)
Previous caesarean section (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 3 (3) | 6 (6)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 10 (10) | 11 (11) | 0 (0) | 0 (0)
Transverse presentation (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Twin pregnancy (Pregnancy, puerperium and perinatal conditions) | 16 (16) | 15 (15) | 0 (0) | 0 (0)
Umbilical cord abnormality (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Umbilical cord around neck (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Umbilical cord prolapse (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Uterine contractions during pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine hypotonus (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Agitation neonatal (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Renal failure neonatal (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervix oedema (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chordee (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian enlargement (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian torsion (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shortened cervix (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Uterine atony (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Apparent life threatening event (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atelectasis neonatal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infantile apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Neonatal hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 13 (13) | 12 (12)
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Neonatal tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Respiratory disorder neonatal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion induced (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Appendicectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Caesarean section (Surgical and medical procedures) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Evacuation of retained products of conception (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Labour induction (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Selective abortion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension neonatal (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypoperfusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocele (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neonatal hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mothers Corifollitropin Alfa 150 µg (N=274) | Mothers recFSH 200 IU (N=267) | Fetuses/Infants Corifollitropin Alfa 150 µg (N=352) | Fetuses/Infants recFSH 200 IU (N=326)
Anaemia (Blood and lymphatic system disorders) | 20 (20) | 17 (17) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 15 (16) | 22 (23) | 2 (2) | 8 (8)
Dyspepsia (Gastrointestinal disorders) | 27 (31) | 22 (23) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (6) | 3 (3) | 16 (16) | 17 (17)
Vomiting (Gastrointestinal disorders) | 20 (22) | 14 (15) | 0 (0) | 3 (3)
Fatigue (General disorders) | 17 (19) | 15 (17) | 0 (0) | 0 (0)
Oedema Peripheral (General disorders) | 21 (26) | 13 (16) | 0 (0) | 0 (0)
Gestational diabetes (Metabolism and nutrition disorders) | 10 (10) | 14 (14) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 25 (28) | 20 (25) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 24 (31) | 31 (37) | 0 (0) | 0 (0)
Antepartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 19 (21) | 14 (19) | 0 (0) | 0 (0)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 22 (22) | 20 (20)
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 18 (18) | 15 (15) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 14 (18) | 10 (16) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 34 (38) | 27 (29) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any scientific paper, presentation, or other communication concerning the clinical trial will first be presented to the Sponsor, at least six weeks ahead of estimated publication or presentation, for written consent. The Sponsor shall have the right to make its consent conditional upon proper representation of the interpretation of both the Sponsor and the investigator(s) in the discussion of the data in such communications.